CLINICAL TRIAL: NCT03719924
Title: Nal-IRI/LV5-FU VERSUS PACLITAXEL AS SECOND-LINE THERAPY IN PATIENTS WITH METASTATIC OESOPHAGEAL SQUAMOUS CELL CARCINOMA A Multi-centre, Randomized, Non-comparative Phase II Study
Brief Title: Nal-iri/lv5-fu Versus Paclitaxel as Second Line Therapy in Patients With Metastatic Oesophageal Squamous Cell Carcinoma
Acronym: OESIRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Shire (Industry); Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 62 - OESIRI
Record Dates: First submitted 2018-09-26; First posted 2018-10-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: ESCC NAL-IRI
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — irinotecan sucrosofate; Paclitaxel

STUDY DESIGN:
Intervention Model Description: All initial characteristics will be described in the overall population and by treatment arm. Evaluation criteria related to efficacy and safety will be described by treatment arm. Initial characteristics of best response and toxicities will be evaluated using usual statistics: for quantitative variables: mean, standard deviation, median, interquartile interval and range and for qualitative variables: frequencies and percentages.
  For the primary evaluation end point, a one-sided 95% confidence interval (CI) will be calculated in the experimental arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A: ONIVYDE (Experimental): ONIVYDE ONIVYDE will be administered first, followed by folinic acid or L-folinic acid and then 5-FU at D1 and D14 ONIVYDE: 70 mg/m² intravenous over 90 minutes Folinic acid: 400 mg/m² intravenous over 30 minutes or L-folinic acid (racemic form L) 200 mg/m² over 30 minutes 5-FU: 2400 mg/m² over 46 hours
  Interventions: Drug: Onivyde
- Arm B: TAXOL (Active Comparator): TAXOL Premedication consists of corticosteroids, H1 antihistamines and H2 antagonists during 30 minutes at time 1 hour before chemotherapy One cycle every 28 days (D1=D28) 80 mg/m2 IV over 60 minutes at D1, D8 and D15
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Onivyde — onivyde will be administered first, followed by folinic acid or L-folinic acid and then 5-FU at D1 and D14.
  Other Names: no other intervention name to add
  Arms: arm A: ONIVYDE
Drug: Paclitaxel — Paclitaxel : 80 mg/m2 IV during 60 minutes at D1, D8 and D15
  Other Names: no other intervention name to add
  Arms: Arm B: TAXOL

SUMMARY:
The aim of our study is to evaluate the efficacy and safety of NALIRI plus 5FU versus paclitaxel as a second-line therapy in patients with locally advanced or metastatic ESCC who had failed to cisplatin- or oxaliplatin-based first-line chemotherapy.

The hypotheses are as follows:

H0: the percentage of patients alive at 9 months of 40% is not useful. H1: the percentage of patients alive at 9 months of 60% is expected.

DETAILED DESCRIPTION:
Principal objective:

• To evaluate the survival of patients at 9 months

Secondary objectives:

* Progression-free survival (PFS) (clinical and/or radiological)
* Overall survival (OS)
* Best response rate during treatment according to RECIST 1.1 criteria (according to the investigator and the centralised review committee)
* Toxicity (NCI CTC 4.0)
* Quality of life (QLQ-C30 and OES18 questionnaires of the EORTC)

Arm A (experimental arm): Nal IRI plus LV5-FU (D1=D28) Nal-IRI: 70 mg/m² intravenous over 90 minutes Followed by intravenous folinic acid 400 mg/m² over 30 minutes or L-folinic acid: 200 mg/m² over 30 minutes And then 5-FU 2,400 mg/m² over 46 hours on D1 to D14

Arm B (control arm): PACLITAXEL (D1=D28) Paclitaxel: 80 mg/m² at D1, D8 and D15

Patients will be randomized in a 1:1 ratio using the minimisation technique. Randomisation will be stratified based on the following factors:

* Centre
* WHO performance status: 0/1 versus 2

An analysis of circulating tumour DNA (using genetic mutations, in particular, TP53, and DNA methylation analyses) will be performed before the 1st cycle of treatment and at D28, in order to look for factors predictive of response to treatment (decrease in unbound DNA).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic oesophageal squamous cell carcinoma
* Patient in failure with 1st-line treatment with oxaliplatin or cisplatin. Patients presenting with resectable disease treated with surgery or neoadjuvant or adjuvant chemotherapy with oxaliplatin or cisplatin (with or without radiotherapy) can be included if a recurrence has occurred less than 6 months after the end of treatment
* Age ≥ 18 years
* Unresectable disease, measurable or not, according to RECIST 1.1 criteria
* WHO performance status ≤ 2
* Neutrophils ≥ 1500/mm3 (without use of haematopoietic growth factors), platelets ≥ 100 000/mm3, haemoglobin ≥ 9 g/dl (blood transfusions are authorised for patients with a haemoglobin less than 9 g/dl)
* Total bilirubin ≤ 2 x ULN (biliary drainage is authorised in case of a biliary obstruction); albumin ≥ 25 g/L; AST ≤ 2.5 x ULN, and ALT ≤ 2.5 x ULN (≤ 5 x ULN in case of hepatic metastases)
* Creatinine clearance ≥ 50 ml/min according to MDRD formula
* A normal ECG or ECG with no clinically significant findings
* Patient able to understand and to sign the informed consent form (or who has a legal guardian able to do so for him/him)
* Women of childbearing potential must have a negative pregnancy blood or urine test within 7 days prior to inclusion
* Women of childbearing potential, as well as men (who have sexual relations with women of childbearing potential) must agree to use an effective method of contraception throughout this study and during the 6 months following administration of the last dose of the study medicinal product
* Patient who is a beneficiary of the Social security system
* Patient for whom regular follow-up is possible.

Exclusion Criteria:

* Known brain or bone metastases
* Clinically significant gastrointestinal disorders, including hepatic, haemorrhagic, inflammatory, obstructive disorders or diarrhoea > grade 1
* History of chronic inflammatory bowel disease
* Gilbert's syndrome
* Interstitial lung disease
* Treatment with St John's Wort
* Medical history of Whipple procedure
* Body mass index < 18.5 kg/m2
* Combination with sorivudine and others analogues as brivudine (irreversibly inhibits the enzyme dihydropyrimidine dehydrogenase)
* History of progressive cancer or in remission of less than 3 years duration (patients who present with a cancer in situ or basal cell or squamous cell skin cancer during the last 3 years are eligible).
* Severe arterial thromboembolic events (myocardial infarction, unstable angina, stroke) less than 3 months before inclusion
* NYHA class III or IV congestive heart failure, ventricular arrhythmia or uncontrolled blood pressure
* Significant neuropathy ≥ grade 2 according to NCI CTCAE criteria (National Cancer Institute Common Terminology Criteria for Adverse Events) v.4.0.
* Known hypersensitivity or allergy to a component of the medicinal products used in the study.
* Known DPD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
survival at 9 months | 9 months
  The principal objective is to evaluate survival at 9 months in patients presenting with metastatic oesophageal squamous cell carcinoma (OSC) treated with Nal-IRI/LV5-FU or with paclitaxel.

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Clinical Progression-free survival and/or radiological Progression free survival will be evaluated
Overall survival (OS) | 1 year
  evaluate the overall survival
Best response rate during treatment | 6 months
  Best response rate during treatment according to RECIST 1.1 criteria (according to the investigator and with centralised review)
Toxicity (NCI-CTC v4) | 6 months
  all observed toxicities, graded according to NCI-CTC v4 and the SAE
Quality of life (questionnaires) | 6 months
  Quality of life (QLQ-C30 questionnaires of EORTC) and OES18 questionnaires of EORTC

CONTACTS AND LOCATIONS:
Overall Officials: DAVID TOUGERON, Principal Investigator — PRODIGE 62 - FFCD 1701
Locations (9):
- France (9):
  - Chu Amiens, Amiens
  - Institut Sainte Catherine, Avignon
  - Hopital Européen, Marseille
  - Ch Le Raincy, Montfermeil
  - Chu Saint Louis, Paris
  - Ch Perpignan, Perpignan
  - Chu de Poitiers, Poitiers
  - Chu Rouen, Rouen
  - Ch Duchenne, St-Malo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Randrian V, Adenis A, Desrame J, Barbier E, Di Fiore F, Lievre A, Dahan L, Laurent-Puig P, Mineur L, Breysacher G, Roquin G, Louafi S, Lopez A, Louvet C, Borg C, Metges JP, Faroux R, Gaba L, Manfredi S, Tougeron D. Nal-IRI/LV5-FU versus paclitaxel as second-line therapy in patients with metastatic esophageal squamous cell carcinoma (OESIRI)-PRODIGE 62: A multicentre, randomised, non-comparative phase II study. Dig Liver Dis. 2020 Mar;52(3):347-350. doi: 10.1016/j.dld.2019.11.014. Epub 2019 Dec 30. PMID 31899122
- [Derived] Tougeron D, Mineur L, Zaanan A, Kadi M, Poisson Ligeza C, Bourgeois V, Martin-Babau J, Fadin A, Jestin le Tallec V, Ly Lebrun V, Dubreuil O, Khemissa Akouz F, Thimonier E, Bouche O, Lievre A, Di Fiore F, Lecomte T, Lepage C, Hautefeuille V; PRODIGE 62-FFCD 1701-OESIRI investigators/collaborators. Nal-IRI/LV5-FU versus paclitaxel as second-line therapy in patients with metastatic esophageal squamous cell carcinoma (PRODIGE 62-FFCD 1701-OESIRI). Eur J Cancer. 2025 Oct 1;228:115741. doi: 10.1016/j.ejca.2025.115741. Epub 2025 Aug 22. PMID 40876084